CLINICAL TRIAL: NCT01055951
Title: Feasibility Study of the Solo™ Insulin Pump
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medingo Ltd (Industry)
Responsible Party: Keren Afek, Medingo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTR-045, VTR-075
Record Dates: First submitted 2010-01-24; First posted 2010-01-26 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Type 1 Diabetes; Insulin Pump Users
Keywords: Insulin pumps; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Solo MicroPump (Experimental)
  Interventions: Device: Solo MicroPump

INTERVENTIONS:
Device: Solo MicroPump — 30 days treatment days with an optional extension period of up to 6 month of treatment.
  Other Names: Solo System

SUMMARY:
The purpose of this study is to assess the safety and usability of the Solo™ insulin MicroPump in subjects with type 1 diabetes who are pump users.

DETAILED DESCRIPTION:
This is a multi center, one arm, open label and prospective study to assess the safety and usability of the Solo™ MicroPump Insulin Delivery System .

The study will include a 30 days treatment period with the Solo MicroPump with no special care required for maintaining glycemic control and with an optional extension period of up to six month.

The study will consist of up to 5 visits and one follow up phone call one week after termination of the study. In case of participating the extension period, additional visits will consist once a month.

Visit 1 includes eligibility, baseline evaluation and training in handling of the Solo™ System. If no additional practice is required patients will be enrolled. Visit 2 will commence and Solo pump will be filled with insulin. If additional practice is required subject will be sent home for an additional training period of a few days practice using saline and then return for visit 2.

Treatment visits will take place at 3, 14 and 30 days after the enrolment. Additional visits will take place at 60, 90 and 180 days depending on the extension period.

Subjects will be asked to record blood glucose measurements, daily activities and carbohydrate consumptions between visits.

Seven days after termination of study treatment a telephone contact with the study subject will take place for the purpose of adverse event reporting and the completion of DTSQ questionnaire.

Measurements that will be used for assessing the safety of the device are glucose levels and any occurrence of AE's.

Subjects will complete DTSQ and Performance questionnaires before and at the end of the treatment period for usability evaluation.

Blood and urine tests will be taken at visit 1 and 5, vital signs and physical examination will be evaluated at all study visits.

ELIGIBILITY:
Inclusion Criteria:

* Age range of:

  * 18 to 60 years in Israel
  * 16 to 60 years in Austria
* Type I diabetes and pump treatment duration of more than 6 months.
* Subjects who are using Humalog®, NovoRapid®, and Apidra® 100U/ml insulin
* Measures glucose at least four times per day.
* No more than one severe hypoglycemic or ketoacidosis episode within one year
* Willing to sign an informed consent.
* Cooperative, willing to attend all study visits.

Exclusion Criteria:

* A1c >= 10.0%
* Two or more documented events of severe hypoglycemia within the previous 12 months
* Diabetes related hospitalization over the past 12 months
* Current significant diabetes-related complications
* Pregnant, lactating or planning to become pregnant during the course of the study
* Substance or alcohol abuse
* Uncontrolled hypertension
* Known dermal hypersensitivity to medical adhesive
* Recurrent episodes of skin infections or dermatological allergies
* Serious or unstable medical or psychological conditions
* Current participation in other clinical studies.
* Working for a competitor company

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Device-related adverse outcome | During treatment period

SECONDARY OUTCOMES:
Mechanical dysfunction and diabetes-related adverse outcome | During treatment period

CONTACTS AND LOCATIONS:
Locations (3):
- Medical University Graz, Gratz, Austria
- Israel (2):
  - Rambam Healthcare Campus, Haifa
  - Sourasky Medical Center, Tel Aviv